CLINICAL TRIAL: NCT02329782
Title: Controlled Evaluation of the Adherence Readiness Program for ART Adherence
Brief Title: Supporting Treatment Adherence Readiness Through Training (START)
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: University of California, Los Angeles (Other); Long Beach Education and Research Consultants (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH104086
Record Dates: First submitted 2014-12-22; First posted 2015-01-01 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: HIV Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ARP intervention (Experimental): Adherence counseling intervention
  Interventions: Behavioral: Adherence Readiness Program
- usual care (No Intervention): no intervention, standard care practices regarding adherence support

INTERVENTIONS:
Behavioral: Adherence Readiness Program — The ARP consists of pre-treatment (including practice trials to determine readiness for and timing of ART initiation), early-treatment, and ongoing maintenance training (using a performance-based, dose regulation mechanism to tailor the amount and intensity) phases
  Arms: ARP intervention

SUMMARY:
Multi-site, randomized controlled trial of the Adherence Readiness Program (ARP) adherence intervention for HIV clients starting or restarting antiretroviral therapy (ART) for the purpose of achieving and sustaining optimal levels of ART adherence and virologic suppression. Eligible participants will be randomized to receive either the ARP intervention or usual care (no intervention) and followed for 24 months.

DETAILED DESCRIPTION:
This study will evaluate the effects of the Adherence Readiness Program (ARP) intervention on the primary outcomes of dose-taking HIV antiretroviral (ART) adherence and undetectable HIV viral load in a multi-site randomized controlled trial. The ARP is based on the Information Motivation Behavioral skills (IMB) model of behavior change and includes (1) brief pill taking practice trials for enhancing pre-treatment adherence counseling and providing a behavioral criterion for determining adherence readiness and the start of treatment, and (2) a performance driven dose regulation mechanism to tailor the amount of counseling (from pre-treatment through the full course of treatment) to the individual needs of the patient and conserve limited resources. Participants will be randomized to receive either the ARP (adherence counseling sessions) or usual care. Primary assessments will be administered at screening and every 6 months after ART initiation over a 24-month follow-up, making it one of the few studies to examine intervention effects longer than one year. Secondary outcomes include dose-timing adherence and CD4 count. If effective, the ARP will provide clinicians with an intervention that (1) informs providers and patients when the patient is ready to adhere well and start treatment, (2) enhances adherence readiness from the outset of treatment through the full course of therapy, and (3) tailors the amount of adherence support based on individual patient need and performance, thus more efficiently using clinic resources, fostering better acceptance from providers and patients, and increasing the likelihood of successful program adoption and dissemination. This emphasis on efficient use of resources will be complemented by a cost-effectiveness analysis to further inform policy decisions regarding the transportability of the intervention and its potential for more wide scale use and sustainability if effective.

ELIGIBILITY:
Inclusion Criteria:

1. The patient's provider views the patient as medically appropriate to begin (ART naïve) or restart ART (has been off ART for at least 2 months), and either

   * plans to start the patient on ART
   * would like to start the patient on ART but the provider or patient is uncertain about the patient's readiness to adhere well.

   Patients who are currently on ART are also eligible if they meet the following criteria, which are specific only to this type of patient:

   i) the patient has 2 or more HIV viral load tests in the past year > 1000 copies/ml ii) the patient has had no HIV viral load tests that were undetectable in the past year iii) the patient has a genotype in the past year that does not show resistance as a reason for virologic failure (detectable viral load) iv) primary care provider views the patient as a good candidate for the study, with the understanding that the patient will interrupt ART if assigned to the intervention.

   Criteria i to iii are intended to define a subgroup of nonadherent patients who are taking very little of their ART medications, as evidenced by the combination of consistently high viral load and no drug resistance. If the patient was taking at least a moderate level of drug and still had consistently high viral load, than they would have evidence of drug resistance. Providers are generally comfortable with this type of patient stopping their medication in order to facilitate the pre-treatment, adherence readiness assessment and training phase of the intervention prior to restarting the patient on treatment.
2. The patient's health status is stable. There is no current acute OI or medical condition that calls for immediate ART, as determined by the patient's provider.
3. Most recent HIV viral load is detectable.
4. If CD4 < 200, the patient is on or will be prescribed prophylactic medication
5. Patient is 18 or older.
6. Patient is able and willing to give informed consent.
7. English speaking.

Exclusion Criteria:

1. Patient just tested HIV+ and their provider suspects the patient may be acutely or recently infected (within past 6 months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
HIV virologic suppression | Month 24
  undetectable HIV viral load at time of assessment
log change in HIV viral load (log change in HIV RNA levels) | Month 24
  log change in HIV RNA levels from baseline to Month 24.
optimal dose-taking adherence (whether at least 85% of prescribed doses were taken) | Month 24
  binary variable representing whether at least 85% of prescribed doses were taken between baseline and Month 24
percent dose-taking adherence | Month 24
  percent of prescribed doses taken between baseline and Month 24
HIV virologic suppression | Month 6
  undetectable HIV viral load at time of assessment
log change in HIV viral load (log change in HIV RNA levels) | Month 6
  log change in HIV RNA levels from baseline to Month 6
optimal dose-taking adherence (whether at least 85% of prescribed doses were taken) | month 6
  binary variable representing whether at least 85% of prescribed doses were taken between baseline and Month 6
percent dose-taking adherence | month 6
  percent of prescribed doses taken between baseline and Month 6

SECONDARY OUTCOMES:
dose-timing adherence | Month 24
  percent of prescribed doses taken within correct time-window between baseline and Month 24
dose-timing adherence | Month 6
  percent of prescribed doses taken within correct time-window between baseline and Month 6
optimal dose-timing adherence | Month 24
  binary variable representing whether at least 85% of prescribed doses were taken within correct time-window between baseline and Month 24
optimal dose-timing adherence | Month 6
  binary variable representing whether at least 85% of prescribed doses were taken within correct time-window between baseline and Month 6
change in CD4 count | Month 24
  change in CD4 count from baseline to Month 24
change in CD4 count | Month 6
  change in CD4 count from baseline to Month 6
clinic attendance (number of missed clinic appointments) | Month 24
  number of missed clinic appointments between baseline and Month 24
clinic attendance (number of missed clinic appointments) | Month 6
  number of missed clinic appointments between baseline and Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Wagner, PhD, Principal Investigator — RAND
Locations (3):
- United States (3):
  - CARE CLinic, Long Beach, California
  - T.H.E. Clinic, Los Angeles, California
  - UCLA Care Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wagner GJ, Seelam R, Hoffman R, Ghosh-Dastidar B. Mediators and moderators of ART adherence effects of supporting treatment adherence readiness through training (START): evidence that START helps vulnerable clients achieve better adherence. AIDS Care. 2022 Oct;34(10):1249-1256. doi: 10.1080/09540121.2021.2006133. Epub 2021 Nov 21. PMID 34802352
- [Derived] Wagner GJ, Hoffman R, Linnemayr S, Schneider S, Ramirez D, Gordon K, Seelam R, Ghosh-Dastidar B. START (Supporting Treatment Adherence Readiness through Training) Improves Both HIV Antiretroviral Adherence and Viral Reduction, and is Cost Effective: Results of a Multi-site Randomized Controlled Trial. AIDS Behav. 2021 Oct;25(10):3159-3171. doi: 10.1007/s10461-021-03188-x. Epub 2021 Apr 2. PMID 33811266
- [Derived] Wagner GJ, Linnemayr S, Ghosh-Dastidar B, Currier JS, Hoffman R, Schneider S. Supporting Treatment Adherence Readiness through Training (START) for patients with HIV on antiretroviral therapy: study protocol for a randomized controlled trial. Trials. 2016 Mar 24;17:162. doi: 10.1186/s13063-016-1287-3. PMID 27009061